CLINICAL TRIAL: NCT03525613
Title: A Phase 3, Multi-Center, Randomized, Double-Masked, Sham-Controlled Study to Compare the Efficacy and Safety of Intravitreal Pegcetacoplan Therapy With Sham Injections in Patients With Geographic Atrophy (GA) Secondary to Age-Related Macular Degeneration (AMD)
Brief Title: A Study to Compare the Efficacy and Safety of Intravitreal APL-2 Therapy With Sham Injections in Patients With Geographic Atrophy (GA) Secondary to Age-Related Macular Degeneration
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Apellis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APL2-304
Record Dates: First submitted 2018-04-20; First posted 2018-05-15 (Actual); Results first posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Geographic Atrophy
MeSH Terms: conditions — Geographic Atrophy | interventions — pegcetacoplan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- APL-2 15mg 0.1 mL Monthly for 24 months (Experimental): A single dose of 15 mg APL-2/0.1 mL will be administered via intravitreal injection in this study. Subjects will receive an injection every month
  Interventions: Drug: APL-2
- APL-2 15mg 0.1 mL EOM for 24 months (Experimental): A single dose of 15 mg APL-2/0.1 mL will be administered via intravitreal injection in this study. Subjects will receive an injection every other month
  Interventions: Drug: APL-2
- Sham Procedure Monthly for 24 months (Experimental): Sham Procedure monthly for 24 months
  Interventions: Other: Sham Procedure
- Sham Procedure Every Other Month for 24 months (Experimental): Sham Procedure every other month for 24 months
  Interventions: Other: Sham Procedure

INTERVENTIONS:
Drug: APL-2 — Complement (C3) Inhibitor
  Other Names: Pegcetacoplan
  Arms: APL-2 15mg 0.1 mL Monthly for 24 months
Drug: APL-2 — Complement (C3) Inhibitor
  Other Names: Pegcetacoplan
  Arms: APL-2 15mg 0.1 mL EOM for 24 months
Other: Sham Procedure — Subjects will receive a Sham procedure every month
  Arms: Sham Procedure Monthly for 24 months
Other: Sham Procedure — Subjects will receive a Sham procedure every other month
  Arms: Sham Procedure Every Other Month for 24 months

SUMMARY:
This is a 24-month, Phase III, multicenter, randomized, double-masked, sham-injection controlled study to assess the efficacy and safety of multiple IVT injections of APL-2 in subjects with GA secondary to AMD.

ELIGIBILITY:
Inclusion Criteria:

The study eye must meet all inclusion criteria. If both eyes meet the inclusion criteria, the eye with the worst visual acuity at the screening visit will be designated as the study eye. If both eyes have the same visual acuity, the right eye will be selected as the study eye.

Ocular- specific inclusion criteria apply to the study eye only, unless otherwise specified.

* Age ≥ 60 years.
* Normal Luminance best corrected visual acuity of 24 letters or better using Early Treatment Diabetic Retinopathy Study (ETDRS) charts (approximately 20/320 Snellen equivalent).
* Clinical diagnosis of GA of the macula secondary to AMD as determined by the Investigator and confirmed by the Reading Center.
* The GA lesion must meet the following criteria as determined by the central reading center's assessment of Fundus Autofluorescence (FAF) imaging at screening:

  * Total GA area must be ≥ 2.5 and ≤ 17.5 mm2 (1 and 7 disk areas [DA] respectively)
  * If GA is multifocal, at least one focal lesion must be ≥ 1.25 mm2 (0.5 DA), with the overall aggregate area of GA, as specified above in 4a.
  * The entire GA lesion must be completely visualized on the macula centered image and must be able to be imaged in its entirety and not contiguous with any areas of peripapillary atrophy.
  * Presence of any pattern of hyperautofluorescence in the junctional zone of GA. Absence of hyperautofluorescence (i.e. pattern = none) is exclusionary.
* Adequate clarity of ocular media, adequate pupillary dilation, and fixation to permit the collection of good quality images as determined by the Investigator.
* Meets the following criteria related to microperimetry:

  * Able to detect fixation target.
  * Total elapsed time to complete the 10-2 68 point exam is ≤ 30 minutes in duration.
  * Reliability test ratio must be ≤ 20%.
  * Subject is willing and able to undertake microperimetry assessment in the opinion of the investigator.
* Female subjects must be:

  * Women of non-child-bearing potential (WONCBP), or
  * Women of child-bearing potential (WOCBP) with a negative pregnancy test at screening and must agree to use protocol defined methods of contraception for the duration of the study and refrain from breastfeeding for the duration of the study.
* Males with female partners of child-bearing potential must agree to use protocol defined methods of contraception and agree to refrain from donating sperm for the duration of the study.
* Willing and able to give informed consent and to comply with the study procedures and assessments.

Exclusion Criteria:

Ocular specific exclusion criteria apply to the study eye only, unless otherwise specified.

* GA secondary to a condition other than AMD such as Stargardt disease, cone rod dystrophy or toxic maculopathies like plaquenil maculopathy in either eye.
* Spherical equivalent of the refractive error demonstrating > 6 diopters of myopia or an axial length >26 mm.
* Any history or active choroidal neovascularization (CNV), associated with AMD or any other cause, including any evidence of retinal pigment epithelium rips or evidence of neovascularization anywhere based on SD-OCT imaging and/or fluorescein angiography as assessed by the Reading Center.
* Presence of an active ocular disease that in the opinion of the Investigator compromises or confounds visual function, including but not limited to, uveitis, other macular diseases (e.g. clinically significant epiretinal membrane (ERM), full thickness macular hole or uncontrolled glaucoma/ocular hypertension. Benign conditions in the opinion of the investigator such as peripheral retina dystrophy are not exclusionary).
* Intraocular surgery (including lens replacement surgery) within 3 months prior to randomization.
* History of laser therapy in the macular region.
* Aphakia or absence of the posterior capsule. Note: YAG laser posterior capsulotomy for posterior capsule opacification done at least 60 days prior to screening is not exclusionary.
* Any ocular condition other than GA secondary to AMD that may require surgery or medical intervention during the study period or, in the opinion of the Investigator, could compromise visual function during the study period.
* Any contraindication to IVT injection including current ocular or periocular infection.
* History of prior intravitreal injection.
* Unable to perform microperimetry reliably in the opinion of the investigator
* Prior participation in another interventional clinical study for intravitreal therapies in either eye (including subjects receiving sham).
* Prior participation in another interventional clinical study for geographic atrophy in either eye including investigational oral medication and placebo.
* Participation in any systemic experimental treatment or any other systemic investigational new drug within 6 weeks or 5 half-lives of the active ingredient (whichever is longer) prior to the start of study treatment. Note: clinical trials solely involving observation, over-the-counter vitamins, supplements, or diets are not exclusionary.
* Medical or psychiatric conditions that, in the opinion of the investigator, make consistent follow-up over the 24-month treatment period unlikely, or would make the subject an unsafe study candidate.
* Any screening laboratory value (hematology, serum chemistry or urinalysis) that in the opinion of the Investigator is clinically significant and not suitable for study participation.
* Known hypersensitivity to fluorescein sodium for injection or hypersensitivity to APL-2 or any of the excipients in APL-2 solution.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 637 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2022-06-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (112):
- United States (67):
  - Arizona Retina & Vitreous Consultants, Phoenix, Arizona
  - California Retina Consultants, Bakersfield, California
  - Retina Vitreous Associates Medical Group, Beverly Hills, California
  - Retinal Diagnostic Center, Campbell, California
  - Retina Consultants of Orange County, Fullerton, California
  - Atlantis Eyecare, Huntington Beach, California
  - University of California, San Diego, Jacobs Retina, La Jolla, California
  - Byers Eye Institute at Stanford, Stanford School of Medicine, Palo Alto, California
  - Doheny Eye Center UCLA, Pasadena, California
  - Retina Consultants San Diego, Poway, California
  - Retinal Consultants Med Group, Inc., Sacramento, California
  - Orange County Retina Medical Group, Santa Ana, California
  - California Retina Consultants, Santa Barbara, California
  - Southwest Retina Research Center, LLC, Durango, Colorado
  - Colorado Retina Associates, Golden, Colorado
  - Retina Group of New England, Waterford, Connecticut
  - Blue Ocean Clinical Research / The Macula Center, Clearwater, Florida
  - National Ophthalmic Research Institute (Retina Consultants of Southwest Florida), Fort Myers, Florida
  - Bascom Palmer Eye Institute, Miami, Florida
  - Bascom Palmer Eye Institute of Naples, Naples, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Southeast Retina Center, PC, Augusta, Georgia
  - Gailey Eye Clinic Retina Center, Bloomington, Illinois
  - Northwestern Feinberg School of Medicine, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Midwest Eye Institute, Indianapolis, Indiana
  - Retina and Vitreous Associates of Kentucky, PSC dba Retina Associates of Kentucky, Lexington, Kentucky
  - Retina Associates New Orleans, Metairie, Louisiana
  - The Retina Care Center, Baltimore, Maryland
  - The Retina Group of Washington, Chevy Chase, Maryland
  - Cumberland Valley Retina Center, Hagerstown, Maryland
  - Mid Atlantic Retina Specialists, Hagerstown, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - New England Retina Consultants, Springfield, Massachusetts
  - Michigan Medicine Kellogg Eye Center, Ann Arbor, Michigan
  - Associated Retinal Consultants, P.C, Grand Rapids, Michigan
  - VitreoRetinal Surgery PA, Minneapolis, Minnesota
  - Sierra Eye Associates, Reno, Nevada
  - Retina Center of NJ, LLC, Bloomfield, New Jersey
  - NJ Retina, Toms River, New Jersey
  - Vision Research Center Eye Associates of NM, Albuquerque, New Mexico
  - Ophthalmic Consultants of Long Island, Lynbrook, New York
  - New York Eye and Ear Infirmary of Mount Sinai, New York, New York
  - Vitreous Retina Macula Consultants of NY, New York, New York
  - Duke University, Duke Eye Center, Durham, North Carolina
  - Research - Retina Vitreous Center, Edmond, Oklahoma
  - Oregon Retina, LLP, Eugene, Oregon
  - Mid Atlantic Retina, Bethlehem, Pennsylvania
  - Retina Vitreous Consultants, Monroeville, Pennsylvania
  - Mid Atlantic Retina, Wills Eye Hospital, Philadelphia, Pennsylvania
  - AIO Visionary Eye Care, West Mifflin, Pennsylvania
  - Charles Retina Institute, Germantown, Tennessee
  - Tennessee Retina, PC, Nashville, Tennessee
  - Retina Research Institute of Texas, Abilene, Texas
  - Texas Retina Associates, Dallas, Texas
  - Houston Eye Associates, Houston, Texas
  - Retina Consultants of Houston, PA, Houston, Texas
  - San Antonia Eye Center, San Antonio, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Retina Associates of South Texas, San Antonio, Texas
  - Retinal Consultants of San Antonio, San Antonio, Texas
  - Brown Retina Institute, San Antonio, Texas
  - Strategic Clinical Research Group, Willow Park, Texas
  - University of Utah - John A. Moran Center, Salt Lake City, Utah
  - Emerson Clinical Research Institute, Falls Church, Virginia
  - University of Wisconsin, Madison, Wisconsin
- Australia (6):
  - Marsden Eye Specialist, Parramatta, New South Wales
  - Adelaide Eye & Retina Clinic, Adelaide, South Australia
  - Save Sight Institute, Sydney, South Block
  - Lions Eye Institute, Nedlands, Western Australia
  - Strathfield Retina Clinic, Strathfield
  - Sydney West Retina, Westmead
- UNIFESP - Federal University, São Paulo, Brazil
- UHN Toronto Western Hospital, Toronto, Ontario, Canada
- Czechia (2):
  - AXON Clinical S.R.O, Prague
  - Gemini Eye Clinic, Zlín
- France (8):
  - CHU Dijon, Bordeaux
  - CHU de Bordeaux, Bordeaux
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Clinique du Val d'Ouest, Écully
  - Hopital Lariboisière, Paris
  - CHNO des Quinze-Vingts, Paris
  - Centre Ophtalmologique d'Imagerie et Laser, Paris
  - CHU de Strasbourg Hopital Civil, Strasbourg
- Germany (8):
  - Universitäts-Augenklinik Bonn, Bonn
  - University Opthalmology Clinic, Freiburg im Breisgau
  - Universitätsmedizin Göttingen Georg-August-Universität, Göttingen
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Augenklinik der LMU München, München
  - Augenzentrum am St. Franziskus-Hospital, Münster
  - Universitäts-Augenklinik, Münster
  - STZ Eyetrial, Tübingen
- Israel (3):
  - Rambam Medical Centre, Haifa
  - Carmel Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
- Italy (3):
  - Ospedale San Raffaele, Milan
  - Luigi Sacco Hospital, Milan
  - IRCCS Fondazione G.B. Bietti, Roma
- Netherlands (2):
  - Academisch Medisch Centrum, Amsterdam
  - Radboud University Medical Center Oogheelkunde, Nijmegen
- Southern Eye Specialists, Christchurch, New Zealand
- Poland (3):
  - Oculomedica Eye Centre, Bydgoszcz
  - Oftalmika Eye Hospital, Bydgoszcz
  - Eye Surgery Center Professor Zagorski, Rzeszów
- Spain (3):
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrir
  - Centro Médico Teknon, Barcelona
  - Centro de Oftalmologia Barraquer, Barcelona
- United Kingdom (4):
  - The Royal Victoria Hospital, Belfast
  - Liverpool University Hospitals NHS Foundation Trust, Liverpool
  - Sunderland Eye Infirmary, Sunderland
  - York Teaching Hospital NHS Foundation Trust, York

REFERENCES:
- [Derived] Sadda S, Hatcher KA, Shah BK, Kondapalli SS, Li C, Baumal CR. Outer Retinal Tubulation and Geographic Atrophy: A Natural History Analysis of Sham Observed Eyes from the OAKS and DERBY Trials. Ophthalmol Ther. 2025 Jul;14(7):1611-1619. doi: 10.1007/s40123-025-01156-5. Epub 2025 May 19. PMID 40388106
- [Derived] Fu DJ, Bagga P, Naik G, Glinton S, Faes L, Liefers B, Lima R, Wignall G, Keane PA, Ioannidou E, Ribeiro Reis AP, McKeown A, Scheibler L, Patel PJ, Moghul I, Pontikos N, Balaskas K. Pegcetacoplan Treatment and Consensus Features of Geographic Atrophy Over 24 Months. JAMA Ophthalmol. 2024 Jun 1;142(6):548-558. doi: 10.1001/jamaophthalmol.2024.1269. PMID 38722644
- [Derived] Heier JS, Lad EM, Holz FG, Rosenfeld PJ, Guymer RH, Boyer D, Grossi F, Baumal CR, Korobelnik JF, Slakter JS, Waheed NK, Metlapally R, Pearce I, Steinle N, Francone AA, Hu A, Lally DR, Deschatelets P, Francois C, Bliss C, Staurenghi G, Mones J, Singh RP, Ribeiro R, Wykoff CC; OAKS and DERBY study investigators. Pegcetacoplan for the treatment of geographic atrophy secondary to age-related macular degeneration (OAKS and DERBY): two multicentre, randomised, double-masked, sham-controlled, phase 3 trials. Lancet. 2023 Oct 21;402(10411):1434-1448. doi: 10.1016/S0140-6736(23)01520-9. PMID 37865470
- [Derived] Tzoumas N, Riding G, Williams MA, Steel DH. Complement inhibitors for age-related macular degeneration. Cochrane Database Syst Rev. 2023 Jun 14;6(6):CD009300. doi: 10.1002/14651858.CD009300.pub3. PMID 37314061

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase III, randomized, double-masked, sham injection-controlled study was conducted in subjects with geographic atrophy (GA) secondary to age-related macular degeneration (AMD) at 110 sites in 13 countries between 31 Aug 2018 and 28 Jun 2022.
Pre-assignment Details: This study consisted of a screening period (up to 30 days), a randomization visit on Day 1, and a treatment period (up to 24 months). Subjects were randomized in a 2:2:1:1 ratio on Day 1 to receive treatment with pegcetacoplan monthly, pegcetacoplan every other month (EOM), sham injection monthly or sham injection EOM, respectively. A total of 637 subjects were enrolled in this study.
Groups:
- Pegcetacoplan Monthly: Subjects received intravitreal (IVT) injections of pegcetacoplan 15 milligram (mg)/0.1 milliliter (mL) once monthly for 24 months.
- Pegcetacoplan EOM: Subjects received IVT injections of pegcetacoplan 15 mg/0.1 mL EOM for 24 months.
- Sham Monthly: Subjects received sham injections once monthly for 24 months. The procedure for sham injection was the same as that used for IVT injection until the actual injection but no actual injection occurred.
- Sham EOM: Subjects received sham injections EOM for 24 months. The procedure for sham injection was the same as that used for IVT injection until the actual injection but no actual injection occurred.
Period: Overall Study
Arm/Group | Pegcetacoplan Monthly | Pegcetacoplan EOM | Sham Monthly | Sham EOM
Started | 213 | 212 | 106 | 106
Completed | 144 | 169 | 76 | 82
Not Completed | 69 | 43 | 30 | 24
Not completed — Adverse Event | 11 | 8 | 3 | 3
Not completed — Lost to Follow-up | 4 | 5 | 3 | 2
Not completed — Physician Decision | 0 | 1 | 0 | 1
Not completed — Consent Withdrawal | 25 | 16 | 12 | 9
Not completed — Death | 20 | 9 | 7 | 1
Not completed — Due to Coronavirus Disease-2019 (COVID-19) impact | 9 | 4 | 5 | 8

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) analysis set included all subjects assigned to treatment.
Groups:
- Pegcetacoplan Monthly: Subjects received IVT injections of pegcetacoplan 15 mg/0.1 mL once monthly for 24 months.
- Sham Pooled: Sham Monthly: Subjects received sham injections once monthly for 24 months.
  Sham EOM: Subjects received sham injections EOM for 24 months.
  The procedure for sham injection was the same as that used for IVT injection until the actual injection but no actual injection occurred.
- Total: Total of all reporting groups
Arm/Group | Pegcetacoplan Monthly | Pegcetacoplan EOM | Sham Pooled | Total
Number analyzed (Participants) | 213 | 212 | 212 | 637
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.0 (7.21) | 78.1 (7.81) | 78.6 (7.20) | 78.6 (7.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 | 122 | 136 | 392
  Male | 79 | 90 | 76 | 245
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 193 | 196 | 193 | 582
  Not Reported | 14 | 12 | 14 | 40
  Unknown | 1 | 3 | 3 | 7
  Asian | 3 | 1 | 2 | 6
  Black or African American | 2 | 0 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 7 | 4 | 16
  Not Hispanic or Latino | 191 | 193 | 192 | 576
  Not Reported | 17 | 12 | 16 | 45
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 152 | 148 | 153 | 453
  France | 15 | 14 | 15 | 44
  Australia | 10 | 14 | 10 | 34
  Germany | 7 | 8 | 11 | 26
  Czechia | 9 | 7 | 5 | 21
  Poland | 6 | 5 | 9 | 20
  United Kingdom | 2 | 5 | 4 | 11
  Italy | 3 | 3 | 3 | 9
  Israel | 3 | 2 | 1 | 6
  Netherlands | 3 | 1 | 0 | 4
  New Zealand | 1 | 2 | 1 | 4
  Spain | 1 | 3 | 0 | 4
  Brazil | 1 | 0 | 0 | 1
GA Lesion Size [fundus autofluorescence (FAF)] in the Study Eye [Mean (Standard Deviation); unit: millimeter square (mm^2)] | 8.2150 (3.91483) | 8.3452 (3.95679) | 8.1581 (3.69739) | 8.2394 (3.85283)

OUTCOME MEASURES:

1. Primary Outcome: Least Squares (LS) Mean Change From Baseline in Total Area of GA Lesions in the Study Eye at Month 12
Description: The GA lesion area was measured by a quantified central reading center based on FAF images. LS mean was calculated using a mixed effect model for repeated measure (MMRM) model. Baseline was defined as the last available, non-missing observation prior to first study drug administration.
Time Frame: Baseline (screening) and Month 12
Population: The modified intent-to-treat (mITT) analysis set included all subjects assigned to treatment who received at least 1 injection of pegcetacoplan or sham and had baseline and at least 1 post-baseline value of GA lesion area in the study eye as assessed by FAF. Subjects with a baseline and at least 1 post-baseline value of the outcome at a scheduled visit by Month 12 were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: mm^2
Arm/Group | Pegcetacoplan Monthly | Pegcetacoplan EOM | Sham Pooled
Number analyzed (Participants) | 202 | 204 | 205
mm^2 | 1.5579 (0.08350) | 1.6512 (0.08118) | 1.9692 (0.08218)
Statistical Analysis 1: Comparison: Pegcetacoplan Monthly vs Sham Pooled; Model included treatment + baseline GA lesion area (<7.5 mm^2 or ≥7.5 mm^2) + analysis visit + presence of choroidal neovascularization (CNV) in the fellow eye (yes or no) + analysis visit × treatment + baseline GA lesion area × analysis visit; Test type: Superiority; p = 0.0004, MMRM model; LS Mean Difference = -0.4114, 95% CI 2-sided [-0.6397 to -0.1831]
Statistical Analysis 2: Comparison: Pegcetacoplan EOM vs Sham Pooled; Model included treatment + baseline GA lesion area (<7.5 mm^2 or ≥7.5 mm^2) + analysis visit + presence of CNV in the fellow eye (yes or no) + analysis visit × treatment + baseline GA lesion area × analysis visit; Test type: Superiority; p = 0.0055, MMRM model; LS Mean Difference = -0.3180, 95% CI 2-sided [-0.5423 to -0.0937]

2. Secondary Outcome: LS Mean Change From Baseline in Total Area of GA Lesions in the Study Eye at Month 24
Description: The GA lesion area was measured by a quantified central reading center based on FAF images. LS mean was calculated using a mixed effect model for repeated measure model. Baseline was defined as the last available, non-missing observation prior to first study drug administration.
Time Frame: Baseline (screening) and Month 24
Population: The mITT analysis set included all subjects assigned to treatment who received at least 1 injection of pegcetacoplan or sham and had baseline and at least 1 post-baseline value of GA lesion area in the study eye as assessed by FAF. Subjects with a baseline and at least 1 post-baseline value of the outcome at a scheduled visit by Month 24 were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: mm^2
Arm/Group | Pegcetacoplan Monthly | Pegcetacoplan EOM | Sham Pooled
Number analyzed (Participants) | 202 | 204 | 206
mm^2 | 3.1237 (0.14327) | 3.2826 (0.13238) | 4.0252 (0.14642)
Statistical Analysis 1: Comparison: Pegcetacoplan Monthly vs Sham Pooled; Model included treatment + baseline GA lesion area (<7.5 mm^2 or ≥7.5 mm^2) + analysis visit + baseline presence of CNV in the fellow eye (yes or no) + analysis visit × treatment + baseline GA lesion area (<7.5 mm^2 or ≥7.5 mm^2) × analysis visit; Test type: Superiority; p < 0.0001, MMRM model; LS Mean Difference = -0.9015, 95% CI 2-sided [-1.3026 to -0.5004]
Statistical Analysis 2: Comparison: Pegcetacoplan EOM vs Sham Pooled; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0002, MMRM model; LS Mean Difference = -0.7426, 95% CI 2-sided [-1.1282 to -0.3570]

3. Secondary Outcome: Mean Change in Total Area of GA Lesions in the Study Eye Through Month 24
Description: The mean change in GA lesion area through Month 24 was measured by assuming a piecewise linear trend in time with knots by FAF images at Months 6, 12, 18, and 24 and was calculated using a MMRM model. Baseline was defined as the last available, non-missing observation prior to first study drug administration.
Time Frame: From Baseline (screening) through Month 24
Population: The mITT analysis set included all subjects assigned to treatment who received at least 1 injection of pegcetacoplan or sham and had baseline and at least 1 post-baseline value of GA lesion area in the study eye as assessed by FAF.
Measure: Mean (Standard Error); unit: mm^2
Arm/Group | Pegcetacoplan Monthly | Pegcetacoplan EOM | Sham Pooled
Number analyzed (Participants) | 202 | 205 | 207
mm^2
  From Baseline to Month 6 | 0.7604 (0.04629) | 0.8220 (0.04346) | 0.9838 (0.04666)
  From Month 6 to Month 12 | 0.7848 (0.05958) | 0.8184 (0.05660) | 0.9710 (0.05163)
  From Month 12 to Month 18 | 0.8004 (0.05034) | 0.8682 (0.04959) | 1.0269 (0.05288)
  From Month 18 to Month 24 | 0.7617 (0.6650) | 0.7499 (0.04372) | 0.9958 (0.05824)
  From Baseline to Month 24 | 3.1073 (0.14841) | 3.2586 (0.13420) | 3.9775 (0.14310)
Statistical Analysis 1: Comparison: Pegcetacoplan Monthly vs Sham Pooled; Estimates for Baseline to Month 6: Model included Treatment + Baseline GA lesion area (< 7.5 mm^2 or >= 7.5 mm^2) + Time (continuous) + Time Spline at Month 6 (continuous) + Time Spline at Month 12 (continuous) + Time Spline at Month 18 (continuous) + Presence of CNV in the fellow eye (Yes or No) + Time (continuous) x Treatment + Time Spline at Month 6 (continuous) x Treatment + Time Spline at Month 12 (continuous) x Treatment + Time Spline at Month 18 (continuous) x Treatment +; Test type: Superiority — Baseline GA lesion area x Time (continuous) + Baseline GA lesion area x Time Spline at Month 6 (continuous) + Baseline GA lesion area x Time Spline at Month 12 (continuous) + Baseline GA lesion area x Time Spline at Month 18 (continuous). A heterogeneous autoregressive covariance matrix was used to model within-subject errors; p = 0.0007, MMRM model; Mean Difference = -0.2234, 95% CI 2-sided [-0.3522 to -0.0946]
Statistical Analysis 2: Comparison: Pegcetacoplan EOM vs Sham Pooled; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.0116, MMRM model; Mean Difference = -0.1618, 95% CI 2-sided [-0.2874 to -0.0361]
Statistical Analysis 3: Comparison: Pegcetacoplan Monthly vs Sham Pooled; Estimates for Month 6 to Month 12: Model included Treatment + Baseline GA lesion area (< 7.5 mm^2 or >= 7.5 mm^2) + Time (continuous) + Time Spline at Month 6 (continuous) + Time Spline at Month 12 (continuous) + Time Spline at Month 18 (continuous) + Presence of CNV in the fellow eye (Yes or No) + Time (continuous) x Treatment + Time Spline at Month 6 (continuous) x Treatment + Time Spline at Month 12 (continuous) x Treatment + Time Spline at Month 18 (continuous) x Treatment +; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.0181, MMRM model; Mean Difference = -0.1862, 95% CI 2-sided [-0.3406 to -0.0318]
Statistical Analysis 4: Comparison: Pegcetacoplan EOM vs Sham Pooled; [analysis description as in outcome 3, analysis 3]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.0467, MMRM model; Mean Difference = -0.1526, 95% CI 2-sided [-0.3030 to -0.0023]
Statistical Analysis 5: Comparison: Pegcetacoplan Monthly vs Sham Pooled; Estimates for Month 12 to Month 18: Model included Treatment + Baseline GA lesion area (< 7.5 mm^2 or >= 7.5 mm^2) + Time (continuous) + Time Spline at Month 6 (continuous) + Time Spline at Month 12 (continuous) + Time Spline at Month 18 (continuous) + Presence of CNV in the fellow eye (Yes or No) + Time (continuous) x Treatment + Time Spline at Month 6 (continuous) x Treatment + Time Spline at Month 12 (continuous) x Treatment + Time Spline at Month 18 (continuous) x Treatment +; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.0019, MMRM model; Mean Difference = -0.2265, 95% CI 2-sided [-0.3696 to -0.0834]
Statistical Analysis 6: Comparison: Pegcetacoplan EOM vs Sham Pooled; [analysis description as in outcome 3, analysis 5]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.0288, MMRM model; Mean Difference = -0.1586, 95% CI 2-sided [-0.3009 to -0.0164]
Statistical Analysis 7: Comparison: Pegcetacoplan Monthly vs Sham Pooled; Estimates for Month 18 to Month 24: Model included Treatment + Baseline GA lesion area (< 7.5 mm^2 or >= 7.5 mm^2) + Time (continuous) + Time Spline at Month 6 (continuous) + Time Spline at Month 12 (continuous) + Time Spline at Month 18 (continuous) + Presence of CNV in the fellow eye (Yes or No) + Time (continuous) x Treatment + Time Spline at Month 6 (continuous) x Treatment + Time Spline at Month 12 (continuous) x Treatment + Time Spline at Month 18 (continuous) x Treatment +; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.0080, MMRM model; Mean Difference = -0.2341, 95% CI 2-sided [-0.4071 to -0.0611]
Statistical Analysis 8: Comparison: Pegcetacoplan EOM vs Sham Pooled; [analysis description as in outcome 3, analysis 7]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.0007, MMRM model; Mean Difference = -0.2459, 95% CI 2-sided [-0.3886 to -0.1031]
Statistical Analysis 9: Comparison: Pegcetacoplan Monthly vs Sham Pooled; Estimates for Baseline to Month 24: Model included Treatment + Baseline GA lesion area (< 7.5 mm^2 or >= 7.5 mm^2) + Time (continuous) + Time Spline at Month 6 (continuous) + Time Spline at Month 12 (continuous) + Time Spline at Month 18 (continuous) + Presence of CNV in the fellow eye (Yes or No) + Time (continuous) x Treatment + Time Spline at Month 6 (continuous) x Treatment + Time Spline at Month 12 (continuous) x Treatment + Time Spline at Month 18 (continuous) x Treatment +; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, MMRM model; Mean Difference = -0.8702, 95% CI 2-sided [-1.2740 to -0.4664]
Statistical Analysis 10: Comparison: Pegcetacoplan EOM vs Sham Pooled; [analysis description as in outcome 3, analysis 9]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.0003, MMRM model; Mean Difference = -0.7189, 95% CI 2-sided [-1.1039 to -0.3339]

4. Secondary Outcome: LS Mean Change From Baseline in Mean Threshold Sensitivity of All Points of the Study Eye at Month 24
Description: Mean threshold sensitivity of all points was determined from the mesopic microperimetry as an assessment of the macular functional response. Microperimetry offers the option to test retinal light sensitivity while directly observing the fundus and allows for monitoring of macular function loss associated with GA progression. The microperimetry reading center overlaid the baseline FAF images with GA lesions traced by the imaging reading center and the corresponding macular integrity assessment microperimetry baseline scanning laser ophthalmoscope image and identified perilesional (within 500 microns outside the atrophy border), paralesional (beyond 500 microns outside the atrophy border), and extralesional (outside the atrophy border) loci on the microperimetry grid to determine the mean threshold sensitivity for these 3 areas. LS mean was calculated using a MMRM model. Baseline was defined as the last available, non-missing observation prior to first study drug administration.
Time Frame: Baseline (screening) and Month 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: decibels (dB)
Arm/Group | Pegcetacoplan Monthly | Pegcetacoplan EOM | Sham Pooled
Number analyzed (Participants) | 179 | 187 | 186
decibels (dB) | -3.319 (0.2969) | -3.064 (0.2331) | -2.954 (0.2156)

5. Secondary Outcome: LS Mean Change From Baseline in Monocular Maximum Reading Speed of the Study Eye at Month 24
Description: The maximum reading speed of the study eye was calculated per Minnesota Low-Vision Reading Test (MNREAD) or Radner Reading Charts user manuals, with no adjustment for reading inaccuracy. An additional step to cap resulting reading speed values at a maximum of 300 words per minute (wpm) was implemented. Maximum reading speed was calculated as the mean of the 3 highest non-zero reading speeds (or 2, or 1 value, as available), except when all wpm were calculated as 0 then the maximum reading speed was calculated as 0. LS mean was calculated using a MMRM model. Baseline was defined as the last available, non-missing observation prior to first study drug administration.
Time Frame: Baseline (screening) and Month 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: wpm
Arm/Group | Pegcetacoplan Monthly | Pegcetacoplan EOM | Sham Pooled
Number analyzed (Participants) | 168 | 181 | 181
wpm | -22.446 (3.0329) | -17.533 (3.2886) | -16.211 (3.8129)

6. Secondary Outcome: LS Mean Change From Baseline in Mean Functional Reading Independence (FRI) Index Score at Month 24
Description: The FRI was an interviewer-administered questionnaire with 7 items on functional reading activities most relevant to GA AMD subjects. It had 1 total index score. For each FRI Index reading activity performed in the past 7 days, subjects were asked about the extent to which they required assistance beyond eyeglasses/contact lenses, including the use of low-vision aids, adjustments in the activity, or help from another subject. Mean FRI Index scores ranged from 1 (unable to do independently) to 4 (totally independent), with higher scores indicating higher functional reading independence. A negative change from baseline indicated a decrease in the FRI; disease worsening. LS mean was calculated using a MMRM model. Baseline was defined as the last available, non-missing observation prior to first study drug administration.
Time Frame: Baseline (screening) and Month 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pegcetacoplan Monthly | Pegcetacoplan EOM | Sham Pooled
Number analyzed (Participants) | 185 | 193 | 195
score on a scale | -0.287 (0.0563) | -0.379 (0.0536) | -0.273 (0.0554)

7. Secondary Outcome: LS Mean Change From Baseline in Normal-Luminance Best-Corrected Visual Acuity (NL-BCVA) Score of the Study Eye at Month 24
Description: The NL-BCVA was assessed by early treatment diabetic retinopathy study (ETDRS) chart prior to dilating the eyes at a starting distance of 4 meters and ranged from 0 (least score) to 100 (best score). If the 4-meter score was >19 letters read correctly, the visual acuity score was the sum of total letters correctly read at 4 meters plus the addition of 30. If the 4-meter score was ≤19 letters read correctly, the visual acuity score was the sum of total letters read correctly at 4 meters and total letters read correctly at the 1-meter distance. If no letters were read correctly at either the 4-meter distance or the 1-meter distance, the visual acuity score was 0. A positive change in the value indicated improvement in visual acuity. LS mean was calculated using a MMRM model. Baseline was defined as the last available, non-missing observation prior to first study drug administration.
Time Frame: Baseline (screening) and Month 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: ETDRS letters score
Arm/Group | Pegcetacoplan Monthly | Pegcetacoplan EOM | Sham Pooled
Number analyzed (Participants) | 202 | 205 | 207
ETDRS letters score | -7.477 (1.0512) | -8.526 (1.0525) | -7.660 (1.0734)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were reported from first study drug administration (Day 1) up to the last visit or early termination visit, 30 days after the last study drug administration for the monthly treatment groups and 60 days after the last study drug administration for the EOM treatment groups, a maximum of 24 months.
Description: The safety analysis set included all subjects randomly assigned to treatment who received at least 1 injection of pegcetacoplan or sham. Ocular TEAEs are presented separately for the study and fellow eyes, and non-ocular (systemic) TEAEs are also presented.
Groups:
- Pegcetacoplan Monthly: Ocular Study Eye: Ocular TEAEs were summarized for the study eye for all subjects who received IVT injections of pegcetacoplan 15 mg/0.1 mL once monthly for 24 months.
- Pegcetacoplan EOM: Ocular Study Eye: Ocular TEAEs were summarized for the study eye for all subjects who received IVT injections of pegcetacoplan 15 mg/0.1 mL EOM for 24 months.
- Sham Pooled: Ocular Study Eye: Ocular TEAEs were summarized for the study eye for all subjects who were randomized to sham monthly and sham EOM treatment groups.
  Sham Monthly: Subjects received sham injections once monthly for 24 months.
  Sham EOM: Subjects received sham injections EOM for 24 months.
  The procedure for sham injection was the same as that used for IVT injection until the actual injection but no actual injection occurred.
- Pegcetacoplan Monthly: Ocular Fellow Eye: Ocular TEAEs were summarized for the fellow eye for all subjects who received IVT injections of pegcetacoplan 15 mg/0.1 mL once monthly for 24 months.
- Pegcetacoplan EOM: Ocular Fellow Eye: Ocular TEAEs were summarized for the fellow eye for all subjects who received IVT injections of pegcetacoplan 15 mg/0.1 mL EOM for 24 months.
- Sham Pooled: Ocular Fellow Eye: Ocular TEAEs were summarized for the fellow eye for all subjects who were randomized to sham monthly and sham EOM treatment groups.
  Sham Monthly: Subjects received sham injections once monthly for 24 months.
  Sham EOM: Subjects received sham injections EOM for 24 months.
  The procedure for sham injection was the same as that used for IVT injection until the actual injection but no actual injection occurred.
- Pegcetacoplan Monthly: Non-ocular: Non-ocular (systemic) TEAEs were summarized for all subjects who received IVT injections of pegcetacoplan 15 mg/0.1 mL once monthly for 24 months.
- Pegcetacoplan EOM: Non-ocular: Non-ocular (systemic) TEAEs were summarized for all subjects who received IVT injections of pegcetacoplan 15 mg/0.1 mL EOM for 24 months.
- Sham Pooled: Non-ocular: Non-ocular (systemic) TEAEs were summarized for all subjects who were randomized to sham monthly and sham EOM treatment groups.
  Sham Monthly: Subjects received sham injections once monthly for 24 months.
  Sham EOM: Subjects received sham injections EOM for 24 months.
  The procedure for sham injection was the same as that used for IVT injection until the actual injection but no actual injection occurred.
Arm/Group | Pegcetacoplan Monthly: Ocular Study Eye | Pegcetacoplan EOM: Ocular Study Eye | Sham Pooled: Ocular Study Eye | Pegcetacoplan Monthly: Ocular Fellow Eye | Pegcetacoplan EOM: Ocular Fellow Eye | Sham Pooled: Ocular Fellow Eye | Pegcetacoplan Monthly: Non-ocular | Pegcetacoplan EOM: Non-ocular | Sham Pooled: Non-ocular
All-Cause Mortality (participants affected / at risk) | 0/213 | 0/212 | 0/211 | 0/213 | 0/212 | 0/211 | 20/213 | 9/212 | 8/211
Serious Adverse Events (participants affected / at risk) | 5/213 | 4/212 | 1/211 | 1/213 | 0/212 | 2/211 | 77/213 | 56/212 | 55/211
Other Adverse Events (participants affected / at risk) | 100/213 | 95/212 | 59/211 | 69/213 | 56/212 | 65/211 | 86/213 | 72/212 | 67/211
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegcetacoplan Monthly: Ocular Study Eye (N=213) | Pegcetacoplan EOM: Ocular Study Eye (N=212) | Sham Pooled: Ocular Study Eye (N=211) | Pegcetacoplan Monthly: Ocular Fellow Eye (N=213) | Pegcetacoplan EOM: Ocular Fellow Eye (N=212) | Sham Pooled: Ocular Fellow Eye (N=211) | Pegcetacoplan Monthly: Non-ocular (N=213) | Pegcetacoplan EOM: Non-ocular (N=212) | Sham Pooled: Non-ocular (N=211)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 1 (1) | 6 (6)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 3 (3) | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papilloedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Disease complication (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endophthalmitis (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 12 (12) | 3 (3) | 3 (4)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 3 (3) | 4 (4)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 4 (5)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Arthritis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blastocystis infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyphaema (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Postoperative thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urethral cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung adenocarcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastases to thorax (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brain stem stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebellar stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intracranial haematoma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intracranial mass (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Genitourinary symptom (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertensive emergency (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Giant cell arteritis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertensive urgency (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegcetacoplan Monthly: Ocular Study Eye (N=213) | Pegcetacoplan EOM: Ocular Study Eye (N=212) | Sham Pooled: Ocular Study Eye (N=211) | Pegcetacoplan Monthly: Ocular Fellow Eye (N=213) | Pegcetacoplan EOM: Ocular Fellow Eye (N=212) | Sham Pooled: Ocular Fellow Eye (N=211) | Pegcetacoplan Monthly: Non-ocular (N=213) | Pegcetacoplan EOM: Non-ocular (N=212) | Sham Pooled: Non-ocular (N=211)
Conjunctival haemorrhage (Eye disorders) | 22 (39) | 19 (25) | 10 (10) | 2 (2) | 3 (3) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 17 (21) | 20 (21) | 17 (28) | 13 (15) | 11 (13) | 19 (25) | 0 (0) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 17 (20) | 19 (25) | 2 (2) | 2 (3) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Neovascular age-related macular degeneration (Eye disorders) | 20 (21) | 14 (15) | 3 (3) | 9 (9) | 5 (5) | 11 (12) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 17 (19) | 16 (18) | 14 (18) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 14 (15) | 14 (15) | 7 (7) | 13 (13) | 13 (14) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Punctate keratitis (Eye disorders) | 16 (16) | 6 (6) | 0 (0) | 9 (9) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitreous detachment (Eye disorders) | 7 (7) | 11 (12) | 8 (8) | 4 (4) | 3 (3) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 4 (4) | 11 (11) | 5 (6) | 3 (3) | 9 (10) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 8 (8) | 4 (5) | 11 (11) | 7 (7) | 6 (6) | 12 (12) | 0 (0) | 0 (0) | 0 (0)
Low luminance best-corrected visual acuity decreased (Eye disorders) | 7 (7) | 5 (5) | 10 (11) | 10 (14) | 6 (7) | 11 (13) | 0 (0) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 9 (10) | 6 (7) | 4 (5) | 10 (15) | 5 (5) | 11 (13) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 23 (26) | 20 (22) | 22 (31)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 15 (16) | 11 (11) | 10 (10)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (11) | 5 (5) | 12 (14)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 16 (17) | 16 (18) | 9 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 15 (21) | 12 (15) | 7 (7)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 12 (15) | 4 (4) | 9 (9)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 20 (20) | 16 (16) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-08-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT03525613/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/13/NCT03525613/SAP_001.pdf